CLINICAL TRIAL: NCT05062629
Title: United States Hypophosphatasia Molecular Research Center
Status: Recruiting | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Eric Rush, Clinical Geneticist, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00001708
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole genome sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Whole Genome Sequencing

SUMMARY:
This study is being done to determine if cryptic alterations exist within or near to the ALPL gene in patients with a clinical diagnosis of hypophosphatasia, but without identifiable alteration on commercial testing. Additionally, the study aims to characterize functional effects of certain variants of uncertain significance in patients with clinical diagnosis of hypophosphatasia.

DETAILED DESCRIPTION:
Primary Study Objectives:

Determine if cryptic alterations exist within or near to the ALPL gene in patients with clinical diagnosis of hypophosphatasia, but without identifiable pathogenic or likely pathogenic variant on commercial testing.

Secondary Study Objective(s):

Characterize functional effects of variants of uncertain significance in patients with clinical diagnosis of hypophosphatasia

Further characterize the differential diagnosis of hypophosphatasemia in patients with skeletal disease

ELIGIBILITY:
Inclusion Criteria:

Aim 1-

1. Diagnosis of Hypophosphatasia based on clinical features that include

   * History consistent with diagnosis of hypophosphatasia AND
   * Physical examination findings consistent with a diagnosis of hypophosphatasia AND
   * Presence of low serum alkaline phosphatase level for age and sex AND
   * Elevation of at least one natural substrate of alkaline phosphatase
2. Lack of detection of a variant on molecular analysis of the ALPL gene. When possible, first degree relatives (parents, siblings, or child) will be included for the sole purpose of trio testing. No additional information will be collected on first degree relatives.

Aim 2-

1. Missense variant in ALPL which is interpreted as a variant of uncertain significance by the American College of Medical Genetics Guidelines for Variant Interpretation
2. Variant has been interpreted as pathogenic, likely pathogenic, likely benign, or benign using ex-US interpretation guidelines

Exclusion Criteria:

Aim 1-

1. History and physical examination incompatible with a diagnosis of hypophosphatasia OR
2. Absence of hypophosphatasemia as measured by age and sex-matched control OR
3. Absence of at least one elevated natural substrate of alkaline phosphatase OR
4. Alternate diagnosis which could overlap with signs and symptoms of hypophosphatasia

Aim 2-

1. Inability to express variant in plasmid for residual enzyme and co-transfection analyses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical diagnosis of hypophosphatasia with negative molecular testing.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of cryptic alterations in the ALPL | 3 years
  Identification of cryptic alterations in the ALPL, with careful focus on cryptic variants within the 12 exons, intronic variants, and variants in regulatory elements.
  Characterization of loss of function or dominant negative effect in variants which are considered to be of uncertain clinical significance by American College of Medical Genetics guidelines for variants interpretation such that variants are able to be reclassified into actionable (pathogenic, likely pathogenic) or nonactionable (benign, likely benign) class

SECONDARY OUTCOMES:
Finding of alternate diagnoses among the cohort of nominated patients | 3 years
  Finding of alternate diagnoses among the cohort of nominated patients, expanding the differential diagnosis of hypophosphatasemia

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rush, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — https://www.childrensmercy.org/childrens-mercy-research-institute/studies-and-trials/hypophosphatasia-molecular-research-center/